CLINICAL TRIAL: NCT02374216
Title: A Prospective Analysis of Failures/Complications With Oral Implants
Brief Title: A Prospective Analysis of Failures of Oral Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Bruno Ramos Chrcanovic, DDS, MSc, PhD student, Malmö University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dnr 2014/333
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Dental Implant Failure; Periodontal Bone Loss
Keywords: Dental Implants; Periodontal Bone Loss; Implant-Supported Dental Prosthesis; Dental Prosthesis Failure
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental implants (Other): Evaluation of the failure rate of all dental implants, of any brand, inserted between September 1st 2014 and August 31st 2017
  Interventions: Procedure: Insertion of dental implants

INTERVENTIONS:
Procedure: Insertion of dental implants — Evaluation of the failure rate of all dental implants, of any brand, inserted between September 1st 2014 to August 31st 2017
  Other Names: Dental implant surgical placement

SUMMARY:
The purpose of this prospective clinical trial is to investigate and identify factors associated with the failure of dental implants within the population rehabilitated with dental implants at the Folktandvården Specialistklinik in Malmö (Spårvägsgatan 12, 214 27, Malmö).

DETAILED DESCRIPTION:
The treatment begins with screening against inclusion and exclusion criteria. The patients will then be informed of the design of the study through the reading of the Form for Patient Information and the Informed Consent in Swedish and verbally.

All dental implants to be inserted will be included in the study. Some surgical, implant, loading, prosthetic variables of the study will be decided according to the surgeon's criteria and patient's decisions.

Data will be collected in specific forms, and will be categorized as surgical, implant-specific, patient-related, anatomic, loading conditions, prosthetic, and complications.

Besides descriptive statistics, Kaplan-Meier analysis will be used to estimate implant survival/failure rates (an estimator for estimating the survival function from lifetime data), and multivariate Cox proportional hazards models will be used to identify prognostic variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a minimum age of 18 years;
* Patients having read, understood, and signed the Form for Patient Information and the Informed Consent.

Exclusion Criteria:

* Age less than 18 years;
* General contraindications for implant surgery;
* Subjects with an untreated systemic disease. A complete medical report will permit the disqualification of subjects with an untreated systemic disease. Patients with a systemic disease such as diabetes or hypertension will not be excluded, as long as these pathologies were treated and stabilized within normal biologic parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Survival of implants | Up to 3 years
  Time from the surgical placement of implants until the last follow-up visit or until its failure

SECONDARY OUTCOMES:
Marginal bone loss | Up to 3 years
  Time from the surgical placement of implants until the last follow-up visit
Dental prosthesis complications | Up to 3 years
  Time from the surgical placement of implants until the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Bruno R Chrcanovic, DDS MSc, Principal Investigator — Malmö University; Ann Wennerberg, DDS PhD, Study Chair — Malmö University; Tomas Albrektsson, MD PhD, Study Chair — Göteborg University / Malmö University; Jenö Kisch, DDS, Study Director — Region Skåne
Locations (1):
- Folktandvården Specialistklinik, Malmo, Skåne County, Sweden